CLINICAL TRIAL: NCT01508624
Title: Evaluation of an Intervention to Increase Pain Relief, Perceived Anxiety and Recovery in Participants Receiving Office Based Surgery
Brief Title: Evaluation of Interventions to Improve Pain Relief, Perceived Anxiety and Recovery in Participants Receiving Office Based Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6045559US
Record Dates: First submitted 2011-12-08; First posted 2012-01-12 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Varicose Veins; Pain
Keywords: Randomised controlled trial; Pain; Recovery; Office based surgery
MeSH Terms: conditions — Varicose Veins; Pain | interventions — Drug Interactions; Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Control (No Intervention): participants will receive standard usual care
- Interaction (Experimental): Participants will interact with nurses during their procedure
  Interventions: Other: Interaction
- Music (Experimental): Participants will listen to music using head phones during their procedure.
  Interventions: Other: Music
- Touch - stress balls (Experimental): Participants will be provided with stress balls to use during their procedure
  Interventions: Behavioral: Touch - stress balls
- DVD (Experimental): Participants will watch a DVD during their procedure and will listen to the accompanying audio through head phones
  Interventions: Behavioral: DVD

INTERVENTIONS:
Other: Interaction — Participants in this condition will interact with nurses during their surgery. The nurses will not touch the patient's hand during treatment as this intervention looks at interaction with another person, in the absence of tactile stimuli.
  Arms: Interaction
Other: Music — Participants will be offered a choice of music to listen to from a selection at the clinic, they will also have the opportunity of bringing or selecting their own music which can be streamed from the internet. They will listen to the music through headphones
  Arms: Music
Behavioral: Touch - stress balls — Participants will be provided with two stress balls which they will be encouraged to squeeze during their surgery and administration of the local anaesthetic
  Arms: Touch - stress balls
Behavioral: DVD — participants will be given a choice of DVDs to watch during their procedure. A wall mounted screen will be positioned so that participants can comfortably view the screen during their procedure. they will listen to the accompanying audio through wireless headphones.
  Arms: DVD

SUMMARY:
This research will evaluate the impact of interventions to improve pain relief and recovery following office based surgery.

There will be three phases to this research. The first phase will focus on predicting recovery from office based vein surgery using a multiple regression analysis.

Phase two will incorporate a randomised controlled trial to compare the effectiveness of a range of interventions in anxiety and pain reduction and recovery for office based vein surgery patients.

The final phase of the investigation will utilise qualitative methodology to explore patients' experiences of each intervention and their opinions about what was and was not effective.

DETAILED DESCRIPTION:
In recent years there has been a large increase in the amount of surgical procedures now available on an outpatient basis (Gilmartin & Wright, 2008). This is due largely to advances in surgical methods and also in response to increasing demands on the National Health Service (M. Mitchell, 2010). This shift impacts patients and health care professionals alike who must adapt to home based recovery and symptom management (Stomberg, Segerdahl, Rawal, Jakobsson, & Brattwall, 2008). This research will investigate patient's expectations, experiences, recovery and satisfaction with office based surgery conducted in a private clinic.

The advancement of office based surgery has led to a rise in the number of procedures completed under local rather than general anaesthetic (Chukmaitov, Devers, Harless, Menachemi, & Brooks, 2011). Resultantly, the number of patients who are conscious during surgery has risen. The environment of the operating theatre must now be considered and nurses are become increasingly responsible for patient's mental wellbeing during surgery. For some, the prospect of being conscious during surgery can be stressful and a number of individual factors have been identified as potentially anxiety provoking (Mitchell, 2009). These range from waiting in the clinic before the surgery (Mitchell, 2008) hearing sounds of instruments being unpacked (Hankela & Kiikkala, 1996) to fears over anaesthesia (Bondy, Sims, Schroeder, Offord, & Narr). Patients' anxiety levels have been found to be high in the pre operative period (Kagan & Bar-Tal, 2008) and the links between high pre operative anxiety and poorer surgical outcomes have been well documented (Dodds 1993,Munafò & Stevenson, 2001).

With this in mind, methods of reducing patient anxiety have been explored. Adapting the operating environment to better suit the needs of the patient has been found to be effective in anxiety reduction (Mark Mitchell, 2008). A powerful yet simple factor in anxiety reduction is the behaviour of the nursing staff in the operating theatre. When nurses use comforting words or touch, anxiety reductions have been observed during and before surgery (Cox & Hayes, 1997.) There is also some evidence to suggest that therapeutic touch can reduce surgical pain(Ramnarine-Singh, 1999). Other easily achievable adaptations to the operating environment that have been shown to have great anti anxiolytic effects include music (Cooke, Chaboyer, & Hiratos, 2005), audio- visual stimuli (Drahota et al., 2008), virtual reality (Hoffman et al, 2001) and massage (Kim, Cho, Woo, & Kim, 2001).

The research above outlines how the addition of fairly minor interventions can be effective in improving patient's experience of office based surgery. As the growth of day surgery continues, identifying and implementing the most effective interventions for anxiety and pain reduction grows ever more important.

In light of the research outlined above, this investigation will utilise a three phase approach t evaluate interventions aimed at improving pain relief and recovery following office based surgery.

ELIGIBILITY:
Inclusion Criteria:

* Participants will need to meet the following inclusion criteria to take part in this research:

  * To be aged over 18,
  * To have given informed consent,
  * To have a good understanding of written and spoken english,
  * To be receiving EVLA or phlebectomies for varicose veins

Exclusion Criteria:

* The following exclusion criteria will be applied:

  * If participants do not wish to take part due to randomisation or intervention procedures
  * If they have a poor understanding of written and spoken english,
  * If they are younger than 18 years of age, or older than 80
  * The presence of leg ulcers
  * If they are having foam treatments for thread veins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2012-04; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Level of pain experienced at the time of surgery | Immediately after surgery, in the recovery area participants will complete a brief measure of pain (The McGill Pain Questionnaire) up to day 1
  Measured by the McGill Pain Questionnaire
Change in pain experienced from time of surgery to 8 weeks after surgery | 8 weeks after date of surgery
  Measured by the McGill Pain Questionnaire

SECONDARY OUTCOMES:
Recovery | 8 weeks
  return to pre surgical functioning, satisfaction with treatment, quality of life, symptom severity,
Anxiety | Immediatley after surgery
  Participants will complete the state scale of the State Trait Anxiety Inventory in the waiting area immediately after surgery to indicate how anxious they felt during their procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Briony Hudson, Principal Investigator — University of Surrey; Jane Ogden, Study Chair — University of Surrey
Locations (2):
- United Kingdom (2):
  - The Whiteley Clinic, Guildford
  - The University of Surrey, Guildford